CLINICAL TRIAL: NCT03203512
Title: Effects of Fish Oil-derived N-3 Polyunsaturated Fatty Acids on the Generation and Functional Activities of Extracellular Vesicles
Brief Title: Fish Oil-derived N-3 Polyunsaturated Fatty Acids and Extracellular Vesicles
Acronym: HI-FIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Principal Investigator, Professor Parveen Yaqoob, MA, DPhil, RNutr, FAfN, Professor Parveen Yaqoob, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: UREC 17/18
Record Dates: First submitted 2017-06-23; First posted 2017-06-29 (Actual); Results first posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Extracellular Vesicles; Generation and Function
Keywords: Fish oil; N-3 polyunsaturated fatty acids
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Fish oil capsules
  Interventions: Dietary Supplement: Fish oil capsules
- Placebo (Placebo Comparator): High-oleic safflower oil capsules
  Interventions: Dietary Supplement: High-oleic safflower oil capsules

INTERVENTIONS:
Dietary Supplement: Fish oil capsules — Each serving contains 360mg eicosapentaenoic acid (EPA), 270mg docosahexaenoic acid (DHA) and total supplement is 1.8 g per day n-3 PUFA for 12 weeks
  Arms: Intervention
Dietary Supplement: High-oleic safflower oil capsules — High-oleic safflower oil capsules for 12 weeks
  Arms: Placebo

SUMMARY:
N-3 polyunsaturated fatty acids (n-3 PUFA), which are abundant in oily fish and fish oils, have been suggested to play a role in reducing the risk of cardiovascular diseases (CVDs) by modifying a wide range of risk factors, such as blood fats, blood clotting, blood vessel function and inflammation. Extracellular vesicles (EVs) are small particles released from various cells when they are activated or damaged. High numbers of EVs in the blood have been associated with a higher risk of CVDs, and it is thought that this is because they carry 'bioactive' components which can affect many processes involved in CVDs. However, very few clinical trials have investigated the relationships between the consumption of n-3 PUFA and circulating EVs. This study aims to investigate the effects of dietary n-3 PUFA on the generation and functional activities of EVs, which would provide new insight into the benefits of n-3 PUFA on cardiovascular health.

DETAILED DESCRIPTION:
The proposed study will be a randomised, double-blind, placebo-controlled crossover intervention. Subjects (40-70y) at moderate CVDs risk will be supplemented with either fish oil (1.8 g/d n-3 PUFA) or placebo (high-oleic safflower oil) for 12 weeks. After a 12-week washout and then cross-over to the other intervention for another 12 weeks. Blood samples will be collected before and after each intervention. A food frequency questionnaire will be administered to assess the subject's habitual intake of n-3 PUFA. Subjects will also be expected to maintain a low consumption of n-3 fatty acids, refrain from the use of all supplements, and maintain their body weight during the study. The dose is based on our previous work, which demonstrated a reduction in numbers of endothelial-derived EVs (EEVs) and a trend for reduced numbers of platelet-derived EVs (PEVs), and a dose at which beneficial effects of n-3 PUFA on plaque stability are reported. The experimental work will follow two main strands. The first strand will examine the influence of n-3 PUFA supplementation on the characteristics and functional activities of total EVs from plasma. The second strand will examine the influence of n-3 PUFA on the generation of PEVs from platelets taken from subjects and stimulated in vitro; the PEVs generated will subsequently be assessed for their composition and functional activity. This experimental design will allow simultaneous investigation of both the composition and activity of total EVs taken directly from blood, and the generation and activity of PEVs. Based on our previous work, 27 subjects are required to detect a 10% reduction in numbers of EVs following fish oil supplementation with a two-sided significance level of 5% and a power of 90%, and 34 subjects are required for a power of 95%. Also based on previous data, 22 subjects would give 95% power to detect 10% differences in thrombus formation and 30 subjects are required to detect a significant effect of n-3 PUFA on platelet aggregation and phosphatidylserine (PS) exposure. Allowing for a 15% dropout rate, and aiming for 95% power based on a 10% reduction in EVs numbers, we will therefore recruit 40 subjects in total.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-70 years
* Non-smoker
* At moderate risk of cardiovascular diseases

  * The risk will be evaluated by an online calculator called "QRISK2". This online calculator (https://qrisk.org/2016/), which use traditional risk factors (age, systolic blood pressure, smoking status and ratio of total serum cholesterol to high-density lipoprotein cholesterol) together with body mass index, ethnicity, measures of deprivation, family history, will provide a percentage of risk of having a heart attack or stroke within the next 10 years.
  * Subjects with 10%-20% will be regarded as being at moderate risk

Exclusion Criteria:

* BMI: <18.5 kg/m2
* Anaemia (haemoglobin concentration <12.5 g/L in men and<11.5 g/L in women)
* Hyperlipidaemia (total cholesterol concentration >8 mmol/L)
* Diabetes (diagnosed or fasting glucose concentration >7 mmol/L) or other endocrine disorders
* Angina, stroke, or any vascular disease in the past 12 months
* Renal, gastrointestinal, respiratory, liver or bowel disease
* Inflammatory disease
* Take drug treatment for hypertension, hyperlipidaemia, inflammation, depression or thyropathy.
* Take aspirin, ibuprofen or other nonsteroidal anti-inflammatory drugs (NSAIDs) > 4 times per month, or once in the week preceding the study
* Take any other anti-platelet or anti-coagulant drugs, like triflusal, clopidogrel and warfarin.
* Have allergies
* Smoking (including e-cigarettes and nicotine products)
* Alcohol misuse or intakes >21 units/wk for men and >15 units/wk for women or have a history of alcohol misuse
* Regularly consume oily fish and/or dietary supplements
* Planning to start or on a weight reducing regimen
* Intense aerobic exercise (>20 min, three times a week)
* Females who are pregnant, lactating, or if of reproductive age and not using a reliable form of contraception (including abstinence)
* Have participated in another clinical trial within the last three months

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parveen Yaqoob, MA, DPhil, RNutr, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, United Kingdom

REFERENCES:
- [Derived] Bozbas E, Zhou R, Soyama S, Allen-Redpath K, Mitchell JL, Fisk HL, Calder PC, Jones C, Gibbins JM, Fischer R, Hester S, Yaqoob P. Dietary n-3 polyunsaturated fatty acids alter the number, fatty acid profile and coagulatory activity of circulating and platelet-derived extracellular vesicles: a randomized, controlled crossover trial. Am J Clin Nutr. 2024 May;119(5):1175-1186. doi: 10.1016/j.ajcnut.2024.03.008. Epub 2024 Mar 13. PMID 38484976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by using the Hugh Sinclair Unit of Human Nutrition volunteer database, emailing advertisements to staff and students of the University of Reading, to members of local community groups and to staff members in large local organisations and companies between Oct 2017 and March 2019. The first participant was enrolled on 16th Feb 2018 and the last participant was enrolled in March 2019.
Pre-assignment Details: Of the 416 participants contacted, a total of 58 participants were screened, of which 14 subjects failed to meet inclusion criteria and 2 declined to participate; 42 participants were enrolled on the trial and 40 completed the study with 2 dropped out before starting.
Groups:
- Fish Oil Capsules, Then Placebo Capsules: Participants received fish oil capsules for in the first 12-week period and after 12-week wash-out, they received placebo capsules for a further 12 weeks
  Fish oil capsules: each serving contains 360mg eicosapentaenoic acid (EPA), 270mg docosahexaenoic acid (DHA) and total supplement is 1.8 g per day n-3 PUFA
  Placebo capsules: high-oleic safflower oil capsules
- Placebo Capsules, Then Fish Oil Capsules: Participants received placebo capsules for in the first 12-week period and after 12-week wash-out, they received fish oil capsules for a further 12 weeks.
  Fish oil capsules: each serving contains 360mg eicosapentaenoic acid (EPA), 270mg docosahexaenoic acid (DHA) and total supplement is 1.8 g per day n-3 PUFA
  Placebo capsules: high-oleic safflower oil capsules
Period: First Intervention (12 Weeks)
Arm/Group | Fish Oil Capsules, Then Placebo Capsules | Placebo Capsules, Then Fish Oil Capsules
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Washout (12 Weeks)
Arm/Group | Fish Oil Capsules, Then Placebo Capsules | Placebo Capsules, Then Fish Oil Capsules
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Second Intervention (12 Weeks)
Arm/Group | Fish Oil Capsules, Then Placebo Capsules | Placebo Capsules, Then Fish Oil Capsules
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fish Oil Capsules, Then Placebo Capsules: Participants received fish oil capsules three times per day with meals for in the first 12-week period and after 12-week wash-out, they received placebo capsules for a further 12 weeks
  Fish oil capsules: each serving contains 360mg eicosapentaenoic acid (EPA), 270mg docosahexaenoic acid (DHA) and total supplement is 1.8 g per day n-3 PUFA
  Placebo capsules: high-oleic safflower oil capsules
- Placebo Capsules, Then Fish Oil Capsules: Participants received placebo capsules three times per day with meals for in the first 12-week period and after 12-week wash-out, they received fish oil capsules for a further 12 weeks.
  Fish oil capsules: each serving contains 360mg eicosapentaenoic acid (EPA), 270mg docosahexaenoic acid (DHA) and total supplement is 1.8 g per day n-3 PUFA
  Placebo capsules: high-oleic safflower oil capsules
- Total: Total of all reporting groups
Arm/Group | Fish Oil Capsules, Then Placebo Capsules | Placebo Capsules, Then Fish Oil Capsules | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.3 [62.8 to 65.8] | 65.0 [62.6 to 66.6] | 65.0 [62.0 to 66.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 16
  Male | 15 | 9 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  White British | 20 | 20 | 40
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 20 | 40
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.0 (2.8) | 25.7 (3.1) | 25.4 (2.9)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 130.5 (11.5) | 137.1 (15.8) | 134.0 (14.2)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 78.5 (7.3) | 79.1 (10.7) | 78.8 (9.1)
Blood Cholesterol Concentration [Mean (Standard Deviation); unit: mmol/L] | 5.8 (0.9) | 6.2 (1.1) | 6.0 (1.0)
Blood Triglyceride Concentration [Median (Inter-Quartile Range); unit: mmol/L] | 1.2 [1.0 to 1.6] | 1.0 [1.0 to 1.5] | 1.2 [1.1 to 1.5]
Blood High Density Lipoprotein Concentration [Median (Inter-Quartile Range); unit: mmol/L] | 1.6 [1.4 to 1.7] | 1.6 [1.5 to 1.7] | 1.6 [1.5 to 1.7]
Blood Glucose Concentration [Mean (Standard Deviation); unit: mmol/L] | 5.9 (0.8) | 5.6 (0.4) | 5.8 (0.6)
10-yr CVD risk (QRISK2) [Mean (Standard Deviation); unit: percentage of risk] — QRISK2, as a scoring system to evaluate cardiovascular risk, includes age, gender, ethnicity, United Kingdom postcode, smoking status, disease information, family history, the ratio of plasma TC to HDL-C, SBP, height and weight, and provides a percentage of risk of having a heart attack or stroke within the next ten years (https://qrisk.org/2017/).
  percentage of risk | 13.0 (0.03) | 12.9 (0.03) | 12.9 (0.03)

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Circulating Total EVs in Platelet-free Plasma (PFP) Detected by Nanoparticle Tracking Analysis (NTA)
Description: Circulating EVs were first isolated to obtain fractions 7~9 by size exclusion chromatography (SEC) using Izon qEV columns (Izon Science Ltd, Oxford, United Kingdom). Fractions were then diluted with PBS to maintain the recommended concentration range of particles (1~10*10^8 vesicles/ml) before being analysed on NanoSight 300 (Malvern, Amesbury, United Kingdom). For each analysis, five videos, each of 60 seconds duration, were captured with the camera level at 13. Data were analysed using the instrument software NTA 3.20, which can identify individual particles and estimate their sizes based on the Stokes-Einstein Equation. Finally, a threshold of 70nm was set for NTA to ensure minimal interference by small lipoproteins.
Time Frame: Change of circulating total EV numbers in PFP detected by NTA after intake period of 12 weeks
Measure: Mean (Standard Error); unit: vesicles per ml blood
Groups:
- Fish Oil Capsules: Participants who received fish oil capsules (1.8 g/d n-3 PUFA) three times per day with meals in either the first or last 12 weeks of the study.
- Placebo Capsules: Participants who received high-oleic safflower oil capsules three times per day with meals in either the first or last 12 weeks of the study.
Arm/Group | Fish Oil Capsules | Placebo Capsules
Number analyzed (Participants) | 40 | 40
vesicles per ml blood | -2.9*10^10 (8.5*10^9) | 7.5*10^9 (4.4*10^9)
Statistical Analysis 1: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of total EV numbers detected by NTA between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on total EV numbers; Test type: Superiority; p < 0.001, ANOVA — Treatment effect: p<0.001; period effect : p=0.552; treatment x period interaction: p=0.622

2. Primary Outcome: Numbers of Total Phosphatidylserine Positive EVs (PS+EVs) in Platelet-free Plasma (PFP) Detected by Flow Cytometry (FCM)
Description: A 5μl of PFP was added into nonsticky microcentrifuge tubes (Alpha Laboratories Ltd, Hampshire, United Kingdom), which contained 5μl FcR blocking reagent (Miltenyi Biotec Ltd, Surrey, United Kingdom) and Annexin V buffer and incubated for 15 minutes in the dark at room temperature. Antibodies and isotype-matched controls were then added and samples incubated for another 15 minutes in the dark at room temperature. After incubation, samples were diluted with 200μl Annexin V buffer and transferred into FACS flow tubes (BD Biosciences, Wokingham, United Kingdom), ready to be analysed by FCM. PS+EVs were identified as Annexin V+EVs when triggering on APC fluorescence.
Time Frame: Change of total PS+EV numbers in PFP detected by FCM after intake period of 12 weeks
Measure: Mean (Standard Error); unit: vesicles per ml blood
Arm/Group | Fish Oil Capsules | Placebo Capsules
Number analyzed (Participants) | 40 | 40
vesicles per ml blood | -1.2*10^7 (2.0*10^6) | -3.0*10^5 (2.5*10^6)
Statistical Analysis 1: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of total PS+EV numbers detected by FCM between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on total PS+EV numbers; Test type: Superiority; p = 0.001, ANOVA — Treatment: p=0.001; period: p=0.646; treatment x period interaction: p=0.267

3. Primary Outcome: Characterisation of Circulating EVs Subpopulation in PFP Detected by Fluorescence FCM
Description: A 5μl of PFP was added into nonsticky microcentrifuge tubes (Alpha Laboratories Ltd, Hampshire, United Kingdom), which contained 5μl FcR blocking reagent (Miltenyi Biotec Ltd, Surrey, United Kingdom) and Annexin V buffer and incubated for 15 minutes in the dark at room temperature. Antibodies and isotype-matched controls were then added and samples incubated for another 15 minutes in the dark at room temperature. After incubation, samples were diluted with 200μl Annexin V buffer and transferred into FACS flow tubes (BD Biosciences, Wokingham, United Kingdom), ready to be analysed by FCM. Platelet-derived EVs (PDEVs) were identified as Annexin V+EVs which also stained positive for CD41-PE in APC vs PE quadrant plot, and endothelial-derived EVs (EDEVs) were identified as Annexin V+EVs which also stained positive for CD105- eFluor450 in APC vs PB quadrant plot.
Time Frame: Change in the numbers of circulating EVs subpopulation in PFP by fluorescence FCM after intake period of 12 weeks
Measure: Mean (Standard Error); unit: vesicles per ml blood
Arm/Group | Fish Oil Capsules | Placebo Capsules
Number analyzed (Participants) | 40 | 40
vesicles per ml blood
  PDEV numbers | -6.0*10^6 (1.5*10^6) | -3.0*10^5 (1.2*10^6)
  EDEV numbers | -5.5*10^5 (1.5*10^5) | 2.9*10^5 (1.3*10^5)
Statistical Analysis 1: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of PDEV numbers detected by FCM between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on PDEV numbers; Test type: Superiority; p = 0.002, ANOVA — Treatment: p=0.002; period: p=0.350; treatment x period interaction: p=0.572
Statistical Analysis 2: Comparison: Fish Oil Capsules vs Placebo Capsules; Test type: Superiority — Null hypothesis is that there was no difference in change of EDEV numbers detected by FCM between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on EDEV numbers; p < 0.001, ANOVA — Treatment: p<0.001; period: p=0.362; treatment x period interaction: p=0.225

4. Secondary Outcome: Pro-thrombotic Activities of Circulating EVs in PFP (Lag Time for Thrombin Generation)
Description: A commercially available, plate-based thrombin generation assay was used to measure thrombin generation in either a standard, pooled vesicle and platelet-free plasma (termed vesicle-free plasma or VFP) or in the same VFP but with added circulating EVs from subjects in the intervention study. This enabled the assessment of TF-dependent thrombin generation specifically attributed to circulating EVs in samples from the intervention study. Results were presented as five variables: (i) lag-phase for initiation of thrombin generation after addition of the trigger (time to 1/6 of the peak height) (min); (ii) peak thrombin concentration (nM); (iii) time to reach the peak (min); (iv) velocity index, defined as = [peak height/(time to peak - lag time)] and (v) area under the curve, defined as endogenous thrombin potential (ETP) (expressed as nM thrombin × min)
Time Frame: Change of pro-thrombotic activities (lag time for thrombin generation)of circulating EVs in PFP after intake period of 12 weeks
Measure: Mean (Standard Error); unit: min
Arm/Group | Fish Oil Capsules | Placebo Capsules
Number analyzed (Participants) | 40 | 40
min | 2.5 (0.5) | 1.2 (0.5)
Statistical Analysis 1: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of EV thrombogenicity in affecting lag time for TF-dependent thrombin generation between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on EV thrombogenicity; Test type: Superiority; p < 0.001, ANOVA — Treatment: p<0.001; period: p=0.010; treatment x period: p=0.608

5. Secondary Outcome: Pro-thrombotic Activities of Circulating EVs in PFP (Peak Thrombin Concentration)
Description: as for outcome 4
Time Frame: Change of pro-thrombotic activities (peak thrombin concentration) of circulating EVs in PFP after intake period of 12 weeks
Measure: Mean (Standard Error); unit: nM
Arm/Group | Fish Oil Capsules | Placebo Capsules
Number analyzed (Participants) | 40 | 40
nM | -16.2 (2.5) | -1.6 (2.0)
Statistical Analysis 1: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of EV thrombogenicity in affecting TF-dependent thrombin peak concentration between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on EV thrombogenicity; Test type: Superiority; p < 0.001, ANOVA — Treatment: p<0.001; period: p=0.073; treatment x period: p=0.667

6. Secondary Outcome: Pro-thrombotic Activities of Circulating EVs in PFP (Time to Peak Thrombin Concentration)
Description: as for outcome 4
Time Frame: Change of pro-thrombotic activities (time to peak thrombin concentration) of circulating EVs in PFP after intake period of 12 weeks
Measure: Mean (Standard Error); unit: min
Arm/Group | Fish Oil Capsules | Placebo Capsules
Number analyzed (Participants) | 40 | 40
min | 4.6 (1.0) | 0.3 (0.7)
Statistical Analysis 1: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of EV thrombogenicity in affecting the time to reach peak TF-dependent thrombin concentration between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on EV thrombogenicity; Test type: Superiority; p < 0.001, ANOVA — Treatment: p<0.001; period: p=0.138; treatment x period: p=0.872

7. Secondary Outcome: Pro-thrombotic Activities of Circulating EVs in PFP (Velocity Index)
Description: as for outcome 4
Time Frame: Change of pro-thrombotic activities (velocity index) of circulating EVs in PFP after intake period of 12 weeks
Measure: Mean (Standard Error); unit: nM/min
Arm/Group | Fish Oil Capsules | Placebo Capsules
Number analyzed (Participants) | 40 | 40
nM/min | -1.1 (0.4) | -0.2 (0.2)
Statistical Analysis 1: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of EV thrombogenicity in affecting TF-dependent velocity index between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on EV thrombogenicity; Test type: Superiority; p = 0.015, ANOVA — Treatment: p=0.015; period: p=0.059; treatment x period: p=0.220

8. Secondary Outcome: Pro-thrombotic Activities of Circulating EVs in PFP (Endogenous Thrombin Potential)
Description: as for outcome 4
Time Frame: Change of pro-thrombotic activities (endogenous thrombin potential) of circulating EVs in PFP after intake period of 12 weeks
Measure: Mean (Standard Error); unit: nM thrombin × min
Arm/Group | Fish Oil Capsules | Placebo Capsules
Number analyzed (Participants) | 40 | 40
nM thrombin × min | -437.2 (70.1) | -60.8 (66.2)
Statistical Analysis 1: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of EV thrombogenicity in affecting TF-dependent endogenous thrombin potential (ETP) between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on EV thrombogenicity; Test type: Superiority; p < 0.001, ANOVA — Treatment: p<0.001; period: p=0.118; treatment x period: p=0.802

9. Secondary Outcome: Ex Vivo Agonist-stimulated Platelet Activation Detected by Plate-based Platelet Aggregation Assay
Description: 96-well high-throughput aggregometry technique, allowing testing of a wide range of concentrations of different agonists, was used to examine the influence of n-3 PUFA supplementation on platelet function. Platelet-rich plasma (PRP) and platelet-poor plasma (PPP) from each study visit was used in the platelet aggregation assay using pre-prepared 96-well microplates, containing the agonists (ADP, EPI, TRAP-6 and U46619). Dose-response curves in response to each agonist were obtained and results were represented as a LogEC50 (log concentration of agonist, M, giving a response halfway between maximum and minimum aggregation).
Time Frame: Change in ex vivo platelet activation after intake period of 12 weeks
Measure: Mean (Standard Error); unit: log(M)
Arm/Group | Placebo Capsules | Fish Oil Capsules
Number analyzed (Participants) | 40 | 40
log(M)
  ADP logEC50 | -0.17 (0.29) | -0.078 (0.11)
  Epinephrine logEC50 | -0.36 (0.24) | 0.16 (0.17)
  TRAP-6 logEC50 | 0.20 (0.18) | 0.058 (0.16)
  U46619 logEC50 | 0.14 (0.30) | -0.37 (0.25)
Statistical Analysis 1: Comparison: Placebo Capsules vs Fish Oil Capsules; Null hypothesis is that there was no difference in change of platelet function in affecting LogEC50 values in response to ADP between fish oil and placebo capsules. Comparisons of this parameter after each intervention were drawn using 2-way ANOVA with the Turkey multiple comparisons test; Test type: Superiority; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Placebo Capsules vs Fish Oil Capsules; Null hypothesis is that there was no difference in change of platelet function in affecting LogEC50 values in response to epinephrine between fish oil and placebo capsules. Comparisons of this parameter after each intervention were drawn using 2-way ANOVA with the Turkey multiple comparisons test; Test type: Superiority; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Placebo Capsules vs Fish Oil Capsules; Null hypothesis is that there was no difference in change of platelet function in affecting LogEC50 values in response to TRAP-6 between fish oil and placebo capsules. Comparisons of this parameter after each intervention were drawn using 2-way ANOVA with the Turkey multiple comparisons test; Test type: Superiority; p > 0.05, ANOVA
Statistical Analysis 4: Comparison: Placebo Capsules vs Fish Oil Capsules; Null hypothesis is that there was no difference in change of platelet function in affecting LogEC50 values in response to U46619 between fish oil and placebo capsules. Comparisons of this parameter after each intervention were drawn using 2-way ANOVA with the Turkey multiple comparisons test; Test type: Superiority; p > 0.05, ANOVA

10. Secondary Outcome: Ex Vivo Agonist-stimulated Platelet Activation Detected by Plate-based Platelet Aggregation Assay (CRP-XL Log EC50)
Description: 96-well high-throughput aggregometry technique, allowing testing of a wide range of concentrations of different agonists, was used to examine the influence of n-3 PUFA supplementation on platelet function. Platelet-rich plasma (PRP) and platelet-poor plasma (PPP) from each study visit was used in the platelet aggregation assay using pre-prepared 96-well microplates, containing the agonists (CRP-XL). Dose-response curves in response to each agonist were obtained and results were represented as a LogEC50 (log concentration of agonist, mg/ml, giving a response halfway between maximum and minimum aggregation).
Time Frame: Change in ex vivo platelet activation after intake period of 12 weeks
Measure: Mean (Standard Error); unit: log (mg/ml)
Arm/Group | Placebo Capsules | Fish Oil Capsules
Number analyzed (Participants) | 40 | 40
log (mg/ml) | -0.39 (0.20) | 0.032 (0.27)
Statistical Analysis 1: Comparison: Placebo Capsules vs Fish Oil Capsules; Null hypothesis is that there was no difference in change of platelet function in affecting LogEC50 values in response to CRP-XL between fish oil and placebo capsules. Comparisons of this parameter after each intervention were drawn using 2-way ANOVA with the Turkey multiple comparisons test; Test type: Superiority; p > 0.05, ANOVA

11. Secondary Outcome: Pro-thrombotic Activities of Platelet-derived Extracellular Vesicles (PDEVs) Prepared From the Supernatants of Stimulated Platelets (Endpoint and Maximum of Thrombus Formation)
Description: Ex vivo thrombus formation was measured by the addition of in vitro-generated PDEVs from stimulated platelets into whole blood under flow. Results were presented as three variables: (i) endpoint for ex vivo thrombus formation (FU); (ii) endpoint for ex vivo thrombus formation (FU); (iii) area under curve.
Time Frame: Change in pro-thrombotic activities (endpoint and maximum of thrombus formation)of PEVs prepared from the supernatants of stimulated platelets after intake period of 12 weeks
Measure: Mean (Standard Error); unit: FU
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 40 | 40
FU
  Endpoint of thrombu formation | -14.3 (13.4) | 9.9 (9.8)
  Maximum of thrombus formation | -1.3 (16.1) | 20.6 (11.1)
Statistical Analysis 1: Comparison: Intervention vs Placebo; Null hypothesis is that there was no difference in change of pro-thrombotic activity of PDEVs in affecting endpoint for ex vivo thrombus formation between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on the pro-thrombotic activity of PDEVs; Test type: Superiority; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Intervention vs Placebo; Null hypothesis is that there was no difference in change of pro-thrombotic activity of PDEVs in affectingamximum for ex vivo thrombus formation between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on the pro-thrombotic activity of PDEVs; Test type: Superiority; p > 0.05, ANOVA

12. Secondary Outcome: Pro-thrombotic Activities of Platelet-derived Extracellular Vesicles (PDEVs) Prepared From the Supernatants of Stimulated Platelets (Area Under Curve)
Description: as for outcome 11
Time Frame: Change in pro-thrombotic activities (area under curve) of PEVs prepared from the supernatants of stimulated platelets after intake period of 12 weeks
Measure: Mean (Standard Error); unit: FU x min
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 40 | 40
FU x min | -945 (4843) | 2502 (3587)
Statistical Analysis 1: Comparison: Intervention vs Placebo; Null hypothesis is that there was no difference in change of pro-thrombotic activity of PDEVs in affecting area under curve for ex vivo thrombus formation between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on the pro-thrombotic activity of PDEVs; Test type: Superiority; p > 0.05, ANOVA

13. Secondary Outcome: Circulating EV Total Lipids Analysis
Description: A 500μl aliquot of frozen PFP was defrosted at room temperature using a roller mixer and subjected to SEC for the isolation and purification of EVs. The fractions 7~9 were pooled together, and 800μl of pooled fractions was prepared for total lipid extraction and methyl esterification. The EV total lipid methyl esters were then analysed by gas chromatography on a Hewlett-Packard 6890 series GC (Hewlett-Packard, California, United States), with the following protocol: split ratio was set as 30:1 for plasma and EV analysis. The injection volume was 1μl for plasma and 5μl for EVs, respectively. The temperature of both injector and detector were kept at 300°C and the temperature program was initial temperature 115°C for 2 minutes, increased at 10 °C/min to 200°C and hold at this temperature for 16 minutes, and finally increased at 60°C/min to 240°C for 2 minutes (total run time: 29.2 minutes). Samples were analysed by using ChemStation software and Microsoft Excel.
Time Frame: Change in total lipids of EVs after intake period of 12 weeks
Measure: Mean (Standard Error); unit: g/100g total fatty acids
Arm/Group | Fish Oil Capsules | Placebo Capsules
Number analyzed (Participants) | 40 | 40
g/100g total fatty acids
  EPA | 0.9 (0.1) | -0.1 (0.1)
  DHA | 1.0 (0.1) | -0.02 (0.1)
  DPA | 0.2 (0.02) | 0.04 (0.03)
  Total n-3 PUFA | 2.5 (0.3) | 0.2 (0.2)
  Oleic acid | -1.9 (0.4) | 0.4 (0.7)
  AA | -0.4 (0.1) | 0.1 (0.1)
  Total MUFA | -2.2 (0.4) | 0.2 (0.8)
Statistical Analysis 1: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of EPA in circulating EV total lipids between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on EPA in circulating EV total lipids; Test type: Superiority; p < 0.001, ANOVA — Treatment: <0.001; period: p=0.978; treatment x period interaction: p=0.140
Statistical Analysis 2: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of DHA in circulating EV total lipids between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on DHA in circulating EV total lipids; Test type: Superiority; p < 0.001, ANOVA — Treatment: p<0.001; period: p=0.699; treatment x period interaction: p=0.114
Statistical Analysis 3: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of oleic acid in circulating EV total lipids between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on oleic acid in circulating EV total lipids; Test type: Superiority; p = 0.011, ANOVA — Treatment: p=0.011; period: p=0.381; treatment x period interaction: p=0.762
Statistical Analysis 4: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of AA in circulating EV total lipids between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on AA in circulating EV total lipids; Test type: Superiority; p < 0.001, ANOVA — Treatment: p<0.001; period: p=0.512; treatment x period interaction: p=0.812
Statistical Analysis 5: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of total n-3 PUFA in circulating EV total lipids between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on total n-3 PUFA in circulating EV total lipids; Test type: Superiority; p < 0.001, ANOVA — Treatment: p<0.001; period: p=0.160; treatment x period interaction: p=0.132
Statistical Analysis 6: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of total MUFA in circulating EV total lipids between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on total MUFA in circulating EV total lipids; Test type: Superiority; p = 0.013, ANOVA — Treatment: p=0.013; period: p=0.500; treatment x period interaction: p=0.522

14. Secondary Outcome: Plasma Total Phospholipids Analysis
Description: A 400μl aliquot of frozen PFP was defrosted and centrifuged to remove denatured protein. The 400μl of 0.9% NaCl was added to the PFP sample to make up 800μl in total, and 30μg of phosphatidylcholine (PC) and 15μg of phosphatidylethanolamine (PE) internal standards were then added for the quantitative analysis. After lipid extraction, separation of PC and PE, and methyl esterification of plasma phospholipid extracts, samples were analysed by GC.
Time Frame: Change of plasma total phospholipids after intake period of 12 weeks
Measure: Mean (Standard Error); unit: g/100g total fatty acids
Arm/Group | Fish Oil Capsules | Placebo Capsules
Number analyzed (Participants) | 40 | 40
g/100g total fatty acids
  EPA | 2.9 (0.2) | -0.1 (0.1)
  DHA | 2.4 (0.2) | -0.1 (0.1)
  DPA | 0.2 (0.04) | -0.1 (0.02)
  Total n-3 PUFA | 5.6 (0.4) | -0.2 (0.1)
  Linoleic acid | -2.0 (0.4) | 0.4 (0.2)
  DGLA | -0.8 (0.1) | 0.04 (0.1)
  Total MUFA | -1.0 (0.4) | -0.1 (0.4)
Statistical Analysis 1: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of EPA in plasma total phospholipids between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on EPA in plasma total phospholipids; Test type: Superiority; p < 0.001, ANOVA — Treatment: p<0.001; period: p=0.169; treatment x period interaction: p=0.629
Statistical Analysis 2: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of DHA in plasma total phospholipids between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on DHA in plasma total phospholipids; Test type: Superiority; p < 0.001, ANOVA — Treatment: p<0.001; period: p=0.262; treatment x period interaction: p=0.150
Statistical Analysis 3: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of DPA in plasma total phospholipids between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on DPA in plasma total phospholipids; Test type: Superiority; p < 0.001, ANOVA — Treatment: p<0.001; period: p=0.302; treatment x period interaction: p=0.385
Statistical Analysis 4: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of linoleic acid in plasma total phospholipids between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on linoleic acid in plasma total phospholipids; Test type: Superiority; p < 0.001, ANOVA — Treatment: p<0.001; period: p=0.793; treatment x period interaction: p=0.522
Statistical Analysis 5: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of dihomo-γ-linolenic acid (DGLA) in plasma total phospholipids between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on DGLA in plasma total phospholipids; Test type: Superiority; p < 0.001, ANOVA — Treatment: p<0.001; period: p=0.956; treatment x period interaction: p=0.238
Statistical Analysis 6: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of AA in plasma total phospholipids between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on AA in plasma total phospholipids; Test type: Superiority; p < 0.001, ANOVA — Treatment: p<0.001; period: p=0.457; treatment x period interaction: p=0.613
Statistical Analysis 7: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of total n-3 PUFA in plasma total phospholipids between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on total n-3 PUFA in plasma total phospholipids; Test type: Superiority; p < 0.001, ANOVA — Treatment: p<0.001; period: p=0.134; treatment x period interaction: p=0.260
Statistical Analysis 8: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of total n-6 PUFA in plasma total phospholipids between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on total n-6 PUFA in plasma total phospholipids; Test type: Superiority; p < 0.001, ANOVA — Treatment: p<0.001; period: p=0.917; treatment x period interaction: p=0.603

15. Secondary Outcome: Concentrations of Lipid Profile in Plasma
Description: A 250μl aliquot of frozen PFP was defrosted at room temperature using a roller mixer and centrifuged at 500xg for 5 minutes at room temperature (Eppendorf Centrifuge 5415 R, DJBlabcare, United Kingdom). Then the sample was analysed by a RANDOX clinical analyser (RANDOX Daytona+ Analyser, Randox Laboratories Ltd, United Kingdom) for the concentration of TC, TAG, HDL-C, LDL-C and TC/HDL-C ratio.
Time Frame: Change in concentrations of plasma lipid profile after intake period of 12 weeks
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Fish Oil Capsules | Placebo Capsules
Number analyzed (Participants) | 40 | 40
mmol/L
  TAG | -0.1 (0.04) | 0.03 (0.04)
  LDL-C | 0.1 (0.06) | -0.1 (0.04)
  TC | 0.1 (0.07) | -0.02 (0.05)
  HDL-C | 0.06 (0.02) | 0.04 (0.02)
  TC/HDL-C ratio | -0.04 (0.05) | -0.1 (0.04)
Statistical Analysis 1: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of plasma TAG between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on plasma TAG; Test type: Superiority; p = 0.016, ANOVA — Treatment: p=0.016; period: p=0.566; treatment x period interaction: p=0.659
Statistical Analysis 2: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of plasma LDL-C between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on plasma LDL-C; Test type: Superiority; p = 0.014, ANOVA — Treatment: p=0.014; period: p=0.842; treatment x period interaction: p=0.943
Statistical Analysis 3: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of plasma TC between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on plasma TC; Test type: Superiority; p = 0.077, ANOVA — Treatment: p=0.077; period: p=0.921; treatment x period interaction: p=0.793
Statistical Analysis 4: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of plasma HDL-C between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on plasma HDL-C; Test type: Superiority; p = 0.379, ANOVA — Treatment: p=0.379; period: p=0.938; treatment x period interaction: p=0.341

16. Secondary Outcome: Concentrations of TC/HDL-C Ratio in Plasma
Description: A 250μl aliquot of frozen PFP was defrosted at room temperature using a roller mixer and centrifuged at 500xg for 5 minutes at room temperature (Eppendorf Centrifuge 5415 R, DJBlabcare, United Kingdom). Then the sample was analysed by a RANDOX clinical analyser (RANDOX Daytona+ Analyser, Randox Laboratories Ltd, United Kingdom) for TC/HDL-C ratio.
Time Frame: Change in concentrations of plasma TC/HDL-C ratio after intake period of 12 weeks
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Fish Oil Capsules | Placebo Capsules
Number analyzed (Participants) | 40 | 40
ratio | -0.04 (0.05) | -0.1 (0.04)
Statistical Analysis 1: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of plasma TC/HDL-C ratio between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on plasma TC/HDL-C ratio; Test type: Superiority; p = 0.285, ANOVA — Treatment: p=0.285; period: p=0.954; treatment x period interaction: p=0.528

17. Secondary Outcome: Blood Pressure
Description: Subjects were asked to have a rest for 10 mins before blood pressure detection, and then blood pressure cuff was placed firmly on their upper left arms approximately 2 cm above the elbow with the indicator mark on the cuff over the brachial artery to start measurement. Subjects should put their arms at the level of the heart and should not speak and cross their legs during the measurement. Measurement was performed three times and waited for 2 mins between each reading ((Omron M2 Upper Arm Blood Pressure Monitor, OMRON Healthcare Europe BV, United Kingdom). The average of the three readings was taken to obtain the final result.
Time Frame: Change in blood pressure after intake period of 12 weeks
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Fish Oil Capsules | Placebo Capsules
Number analyzed (Participants) | 40 | 40
mmHg
  SBP | -6.7 (1.0) | 3.4 (1.7)
  DBP | -2.9 (0.7) | 0.9 (0.9)
Statistical Analysis 1: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of SBP between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on SBP; Test type: Superiority; p < 0.001, ANOVA — Treatment: p<0.001; period effect: p=0.011; treatment x period interaction: p=0.033
Statistical Analysis 2: Comparison: Fish Oil Capsules vs Placebo Capsules; Null hypothesis is that there was no difference in change of DBP between fish oil and placebo capsules. A general linear model with fixed factors of treatment and period was conducted to determine the differences in the effect of two treatments and two periods on DBP; Test type: Superiority; p = 0.002, ANOVA — Treatment: p=0.002; period: p=0.952; treatment x period interaction: p=0.114

ADVERSE EVENTS:
Time Frame: 9 months
Groups:
- Fish Oil Capsules: Participants received fish oil capsules for in the first 12-week period.
  Fish oil capsules: each serving contains 360mg eicosapentaenoic acid (EPA), 270mg docosahexaenoic acid (DHA) and total supplement is 1.8 g per day n-3 PUFA.
- Placebo Capsules: Participants received placebo capsules for in the first 12-week period.
  Placebo capsules: high-oleic safflower oil capsules
Arm/Group | Fish Oil Capsules | Placebo Capsules
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 1/40 | 0/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fish Oil Capsules (N=40) | Placebo Capsules (N=40)
Lump above the site of venepuncture (General disorders) | 1 (1) | 0 (0) — RM Venepuncture left arm - lump above the site (crease of the elbow). localized swelling, no signs of bruising, redness or warmth. This adverse event only happened once during the first arm (when he were taking fish oil capsules firstly)

LIMITATIONS AND CAVEATS:
The collection, isolation and characterization of EVs are still undergoing standardization, so although the protocol for the characterization of EVs applied in this study was refined by combining NTA and fluorescence FCM, circulating EVs measured in this study did not represent all types of EVs as neither NTA nor FCM was able to provide a full picture of the EV population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT03203512/Prot_SAP_000.pdf